CLINICAL TRIAL: NCT01790204
Title: A Study of the Effects of PEITC on Oral Cells With Mutant p53
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R01CA1000853
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2013-11

CONDITIONS: Oral Cancer
Keywords: mutant p53; watercress; Phenethyl isothyocyanate; oral cells of smokers
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Watercress Juice (Experimental): The juice is prepared, by a trained member of the Chung laboratory staff, in the following manner; each serving of watercress juice will be prepared with 55gm watercress (from a local grocery store) with 220 ml purified water, for a proportion of 1:4 (w/w). The watercress and water will be placed in a 1.5 L mechanical blender and blended at low speed for approximately 15 seconds, followed by blending at a high speed for one additional minute. The resulting suspension will be filtered through two layers of cheese cloth. Remaining liquids will be manually extracted from the cheese cloth into the same container. Each serving will be measured to 200 ml. The remaining 20 ml will be used for analysis of ITC content. Each serving will be prepared and kept at 40 C until needed, no more than one hour prior to participant consumption by the subject.
  Interventions: Dietary Supplement: Watercress Juice

INTERVENTIONS:
Dietary Supplement: Watercress Juice — The juice is prepared, by a trained member of the Chung laboratory staff, in the following manner; each serving of watercress juice will be prepared with 55gm watercress (from a local grocery store) with 220 ml purified water, for a proportion of 1:4 (w/w). The watercress and water will be placed in a 1.5 L mechanical blender and blended at low speed for approximately 15 seconds, followed by blending at a high speed for one additional minute. The resulting suspension will be filtered through two layers of cheese cloth. Remaining liquids will be manually extracted from the cheese cloth into the same container. Each serving will be measured to 200 ml. The remaining 20 ml will be used for analysis of ITC content. Each serving will be prepared and kept at 40 C until needed, no more than one hour prior to participant consumption by the subject.

SUMMARY:
The aim of this clinical trial is to examine the effects of phenethyl isothiocyanate (PEITC), a compound derived from cruciferous vegetables, on oral cells with mutant p53. The p53 protein's normal (wild-type) function within cells is to act as a tumor suppressor, or anti-cancer protein. When mutated, the p53 protein not only no longer executes the functions of a tumor suppressor, and it can gain functions as a pro-cancer protein.22 The proposed clinical trial will utilize oral cells collected from subjects who are heavy smokers. Since the subjects are regularly exposed to mutagenic chemicals it is the thought that their oral cells will contain measurable levels of mutant p53. The participants will consume watercress juice, which is rich in PEITC (See Figure 1). Previous studies in the laboratory showed PEITC selectively depletes mutant p53, and not wild type p53, in cell culture. Our hypothesis is that the ITC in the watercress juice will lead to the depletion of mutant p53 within the oral cells. This depletion could lead to a possible clinical application of this compound, such as chemopreventives or oncologic treatments of individuals with oral cancers.

ELIGIBILITY:
Inclusion Criteria:

* Heavy Smoker
* Between the ages of 20 and 65
* Must be able to show proof of citizenship or residency of the United States
* Able to sign and understand a standard consent form

Exclusion Criteria:

* Pregnant or Breast-feeding
* Having any of the following medical conditions:
* Leukoplakia
* Oral Lesions
* Cancer
* Any oral disease that causes sores, ulcerations, irritations, etc.
* Stomach or Intestinal Ulcers
* IBS (Irritable Bowel Syndrome)
* Kidney Disease
* Allergies to watercress or other Cruciferous Vegetables
* Strict Vegetarians or Vegans
* Religious Consumers of Watercress or other Cruciferous Vegetable Juices
* On any of the following medications:
* Chlorzoxazone (Parafon Forte, Paraflex)
* Lithium
* Water Pills/Diuretics (Thiazide or Lasix)
* Warfarin (Coumadin)
* Vitamin K supplements
* H2 acid blocker (Zantac, Pepcid, Axid, Tagamet)
* Proton Pump Inhibitor (Prevacid)
* Digoxin
* Antibiotics
* Diabetic Medications (Insulin)
* Inhaled Bronchodilator
* Oral Steroids (Prednisone, Medrol)
* Inhaled Steroids (Flonase)
* Raloxifene or Tamoxifen
* Thyroid Hormone Replacement

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Evidence of reduced number of oral cells with mutant p53 after administration of PEITC derived from watercress, a cruciferous vegetable. | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Fung-Lung Chung, Ph.D., Principal Investigator — Lombardi Comprehensive Cancer Center
Locations (1):
- Georgetown Clinical Research Unit, Washington D.C., District of Columbia, United States